CLINICAL TRIAL: NCT03296384
Title: Influence of Environmental Factors on the Prevalence, Risk and the Clinical Manifestations of Schizophrenia
Brief Title: Influence of Environmental Factors and Schizophrenia
Acronym: Envschi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut national d'étude démographique (INED) (Unknown); CPN (INSERM U894) CH Sainte-Anne - Paris (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Fondation FondaMental (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P100134
Record Dates: First submitted 2016-09-01; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Patients With Schizophrenia; Relatives
Keywords: schizophrenia; environmental factors
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with schizophrenia (Other)
  Interventions: Other: Clinical and environmental evaluation
- Relatives (Other)
  Interventions: Other: Clinical and environmental evaluation

INTERVENTIONS:
Other: Clinical and environmental evaluation — For schizophrenic's patients, specific assessment will be perform

SUMMARY:
Schizophrenia is a chronic and severe mental disorder with a lifetime prevalence of about 1 per cent, the symptoms can be very disabling and causing a heavy medical and socioeconomic.

There are significant variations from one population to another. Clinical manifestations of schizophrenia (symptoms, evolution, severity of disability) are highly variable. This variability, both epidemiological and clinical, is due to genetic and environmental factors.

Environmental factors may be either risk factors or modifying factors (changing clinical presentation but do not alter the risk of disease) for schizophrenia.

Environmental risk factors have been identified (eg: urbanity, cannabis, migration), but the investigators don't know neither the components directly responsible, nor the mechanisms by which they increase the risk of schizophrenia.

To date, there is no study has systematically evaluated the role of environmental modifying factors in schizophrenia.

Environmental factors may be individual, unique to each person (eg cannabis, migration.), or population-based (eg ethnic density, socio-economic difficulties.) The identification/ identifying of environmental risk factors or modifiers, both individual and population, may have theoretical implications (understanding of etiopathogenic mechanisms) and practical (implementation of preventive measures). The potential effectiveness of preventive measures is even greater than the risk attributable to certain environmental factors is important.

Most studies on environmental factors in schizophrenia were conducted in Anglo-Saxon countries and northern Europe, but no study of these risk factors has been conducted in France.

There are important differences environment based on study populations, these results are not generalizable to other countries, including France.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Age > 18 years
* Somatic state / condition and level of understanding (language, intellectual level) compatible with the data collection (interview, self-administered questionnaires)

Patients

* Diagnosis of schizophrenia according to DSM-IV criteria
* Living in catchment areas

Non-Inclusion Criteria:

All subjects

* Not affiliated to the social security scheme
* inability to provide informed consent
* Decompensated schizophrenic underway

Relatives

* Protective Measures (tutor, curator)

Exclusion criteria:

Patients

* The diagnosis of psychotic disorder is not confirmed by the synthesis of all clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The prevalence of schizophrenia (according to Diagnostic and Statistical Manual of Mental Disorders (DSM IV)) will be estimated from the census population-unit (unit TRIRIS INSEE) | 56 months, From March 2014 to November 2018
The frequency of populational risk factors (insecurity, disorganization and density of migrants) will be assessed from the variables of INSEE | 56 months, From March 2014 to November 2018

SECONDARY OUTCOMES:
The frequency of individual risk factors (migration, cannabis, seasonality of birth, childhood trauma, social environment) will be measured from standardized assessments | 56 months, From March 2014 to November 2018

CONTACTS AND LOCATIONS:
Overall Officials: Franck Schürhoff, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pierre-Michel Llorca, MD PhD, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- Henri Mondor Hospital, Créteil, France